CLINICAL TRIAL: NCT04269928
Title: An Parallel Control Clinical Trail on Effects of Adrenal Artery Ablation and Adrenalectomy in Patients With Primary Aldosteronism
Brief Title: Effects of Adrenal Artery Ablation and Adrenalectomy in Patients With Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Other Study IDs: Quadruple A -PA
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Primary Aldosteronism; Hypertension
Keywords: Primary Aldosteronism; Hypertension; Adrenal Artery Ablation; Adrenalectomy
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adrenal Artery Ablation: Patients in the intervention group will be treated with ablation of adrenal gland by endovascular injection of dehydrated alcohol
  Interventions: Procedure: Endovascular chemical ablation of adrenal gland
- Adrenalectomy: Patients in this group will be treated with unilateral laparoscopic adrenalectomy

INTERVENTIONS:
Procedure: Endovascular chemical ablation of adrenal gland — Patients in this group will be treated with ablation of adrenal gland by endovascular injection of dehydrated alcohol
  Groups: Adrenal Artery Ablation

SUMMARY:
Primary aldosteronism (PA) is the main cause of secondary hypertension, affecting 5-15% of the general hypertensive population. Early diagnosis and treatment are of crucial importance as patients with PA are more susceptible to cardiovascular and cerebrovascular morbidity and mortality than blood-pressure-matched hypertensive patients.

Current guidelines indicate that mineralocorticoid receptor (MR) antagonists and laparoscopic adrenalectomy are the principal treatments for PA.Laparoscopic adrenalectomy is recommended for patients with aldosteronoma or unilateral adrenal hyperplasia. During the past two decades, catheter-based arterial embolization or computed tomography (CT)-guided radiofrequency thermogenesis have been used for aldosteronomas treatment. Although these procedures are claimed to be effective for treatment of aldosteronomas, the evidence comes mostly from case reports or small series. In addition, some PA patients refuse surgery and are intolerant of the adverse effects of MR antagonists; others have persistence of PA after adrenelectomy, but respond poorly to MR antagonists. An alternative therapy is needed in such cases.

In recent years, adrenal artery ablation has also been used to treat primary aldosteronism, which can reduce the level of aldosterone and blood pressure, but its efficacy and safety are not clear. To confirm the effect of adrenal artery ablation on blood pressure, RAAS system and blood potassium, the researchers conducted a parallel control clinical study of patients with primary aldosteronism (Aldosteronoma).

ELIGIBILITY:
Inclusion Criteria:

* Primary aldosteronis diagnosed by increased aldosterone-to-renin ratio (ARR) and serum aldosterone levels ≥15 ng / dl, and confirmed by saline injection test or captopril inhibition test.
* Aldosteronoma had lateralization by adrenal venous sampling (AVS) and confirmed with CT
* Signed informed consent and agreed to participate in this study.

Exclusion Criteria:

* Aldosterone cancer.
* Hyperkalemia.
* Renal failure or the following history of nephropathy: serum creatinine 1.5 times higher than the upper limit; dialysis history; or nephrotic syndrome.
* Secondary hypertension except the primary aldosteronism.
* Adrenergic insufficiency.
* Heart failure with NYHA Ⅱ-Ⅳ grade or unstable angina, severe cardiovascular and cerebrovascular stenosis, myocardial infarction, intracranial aneurysm, stroke and other acute cardiovascular events.
* Acute infections, tumors and severe arrhythmias, psychiatric disorders, drugs or alcohol addicts.
* Liver dysfunction or the following history of liver disease: AST or ALT 2 times higher than the upper limit, liver cirrhosis, history of hepatic encephalopathy, esophageal variceal history or portal shunt history.
* Coagulation dysfunction.
* Pregnant women or lactating women.
* Participated in other clinical trials or admitted with other research drugs within 3 months prior to the trial.
* Allergy or any contraindications for contrast agents and alcohol.
* Refused to sign informed consent

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change of office systolic and diastolic pressure | 52 weeks (End of Trial)
  Change of office systolic and diastolic pressure between the intervention and control group at the end of the study (24 weeks)

SECONDARY OUTCOMES:
Change of 24-h average systolic blood pressure | 52 weeks (End of Trial)
  Change of 24-h average systolic blood pressure between the intervention and control group at the end of the study (24 weeks)
Change of 24-h average diastolic blood pressure | 52 weeks (End of Trial)
  Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure between the intervention and control group at the end of the study (24 weeks)
Change of home systolic and diastolic pressure | 52 weeks (End of Trial)
  Change of home systolic and diastolic pressure between the intervention and control group at the end of the study (24 weeks)
Change of anti-hypertensive regimen | 52 weeks (End of Trial)
  Change of number, classes, and combinations of classes of antihypertensive drugs between the intervention and control group at the end of the study (24 weeks)
Change of blood electrolytes（serum potassium and natrium in mmol/L） | 52 weeks (End of Trial)
  Change of blood electrolytes（serum potassium and natrium in mmol/L）compared with baseline, and between the intervention and control group at the end of the study (24 weeks)between the intervention and control group at the end of the study (24 weeks)
Change of aldosterone-to-renin ratio (ARR） | 52 weeks (End of Trial)
  Change of aldosterone-to-renin ratio (ARR）compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of plasma aldosterone | 52 weeks (End of Trial)
  Change of plasma aldosterone compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of plasma renin | 52 weeks (End of Trial)
  Change of plasma renin compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of plasma cortisol | 52 weeks (End of Trial)
  Change of plasma cortisol compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of serum creatinine | 52 weeks (End of Trial)
  Change of serum creatinine compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of estimated glomerular filtration rate(eGFR) | 52 weeks (End of Trial)
  Change of estimated glomerular filtration rate(eGFR) compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of 24-h urine microalbumin, microalbumin/creatinine ratio | 52 weeks (End of Trial)
  Change of 24-h urine microalbumin, microalbumin/creatinine ratio compared with baseline, and between the intervention and control group at the end of the study (24 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No